CLINICAL TRIAL: NCT03789071
Title: Evaluation of Upper Airway Ultrasound-derived Indexes as Predictors of Difficult Airway
Brief Title: Ultrasound to Predict Difficult Airway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor. Department of Anesthesiology, Augusta University
Other Study IDs: 1218610
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient scheduled for general anesthesia with intubation: Patients in this group (only group) will have clinical airway assessment and external ultrasound assessment of the airway
  Interventions: Diagnostic Test: External ultrasound evaluation of the airway

INTERVENTIONS:
Diagnostic Test: External ultrasound evaluation of the airway — Patients scheduled to have surgery under general anesthesia in whom tracheal intubation is planned, will have a clinical and ultrasound assessment of the airway before surgery. Information regarding laryngoscopy in the operating room will be recorded.

SUMMARY:
Upper airway ultrasound is a valuable, non-invasive, simple, and portable point of care tool for evaluation of the airway, even in the presence of anatomic distortion caused by pathology or trauma. The ultrasound technology is being increasingly adopted in modern anesthesiology practice. As early as in 1984, some authors have recommended its use to guide venous cannulation, because it shortens procedural times, reduces the number of failed puncture attempts, and minimizes complications. On the other hand, ultrasound-guided techniques are considered the gold standard for peripheral nerve blocks.

As ultrasound becomes more widespread, it is important to for anesthesiologists to be aware of the expanding applications of this technology. Current and potential future applications of ultrasound in anesthesiology are wide and include regional anesthesia, neuraxial and chronic pain procedures, vascular access, airway assessment, lung ultrasound, ultrasound neuro-monitoring, gastric ultrasound, focused transthoracic echography, trans-esophageal echocardiography and vascular Doppler flow assessment. The major disadvantage is inter-observer variability, and the fact that it requires is a unique skill that requires continuing training and experience to master the technology. In order to be successful with this technique, it is important to develop a thorough understanding of the sonoanatomy. The normal or abnormal structures need to be imaged and interpreted before any intervention.

Airway management is one of the most important tasks for anesthesiologists. Access to the airway should be safe, fast and efficient. Appropriate planning is crucial to avoid morbidity and mortality when difficulty is anticipated. Inability to maintain airway ventilation is a life-threatening situation that may warrant emergent surgical access to prevent devastating consequences. A thorough assessment of the airway is recommended to predict difficulty. Multiple clinical predictors have been used in clinical practice; however, most of them are associated with low predictive values. In consequence, a comprehensive airway examination that incorporates both quantitative and qualitative tests increases the probability of predicting difficult intubation. Regardless of the method of airway evaluation, it is important to acknowledge that clinical airway assessment is not fully accurate and can produce both false-negative and false-positive results.

There is a growing academic interest in the ability of ultrasound to determine airway size to estimate appropriate endotracheal tube size. Ultrasound enables us to identify important sonoanatomy of the upper airway including thyroid cartilage, epiglottis, cricoid cartilage, cricothyroid membrane, tracheal cartilages, and esophagus. Transverse and parasagittal views can help diagnose supraglottic, glottic and infraglottic airway conditions and aid the anesthesiologist in airway management. Ultrasonography has brought a paradigm shift in the practice of airway management. With increasing awareness, portability, accessibility and further sophistication in technology, it is likely to find a place in routine airway management.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Age older than 18 years

Exclusion Criteria:

* Emergency surgery
* Nasal intubation
* Intubation with fiberoptic scope or glidescope
* Intubation without laryngoscopy
* Awake intubation
* Allergy to ultrasound gel

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for elective surgery under general anesthesia in whom tracheal intubation is planned.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound depth of the tongue | 10 minutes
  With curvilinear ultrasound probe in longitudinal position over upper neck, the distance from probe to tongue will be measured.
Degree of glottic visualization | 10 minutes
  During laryngoscopy, percentage of glottic opening will be recorded

SECONDARY OUTCOMES:
Ultrasound depth of cricoid cartilage | 10 minutes
  With curvilinear ultrasound probe in longitudinal position over upper neck, the distance from probe to the cricoid cartilage will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided